CLINICAL TRIAL: NCT01377896
Title: The Purpose of the Study is to Gain an In-depth Picture of the Patient Management and Prescription Behaviours
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-NZA-XXX-2011/1
Record Dates: First submitted 2011-06-14; First posted 2011-06-22 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Schizophrenia; Bipolar Disorders; Major Depressive Disorders
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
'Real life' retrospective patient cases (10) to provide an objective and robust analytical report of patient management and prescriptions behaviours for Schizophrenia, Bipolar disorders and Major depressive disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with one of the following conditions: Schizophrenia, Bipolar disorders and Major depressive disorders.

Exclusion Criteria:

* Patients who have not been diagnosed with the conditions as outlined in the Inclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cardiovascular events
Sampling Method: Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)